CLINICAL TRIAL: NCT01689740
Title: A Randomized, Double-Blind, Active Placebo-Controlled Phase 2 Pilot Study of MDMA-assisted Psychotherapy in People With Chronic, Treatment-Resistant Posttraumatic Stress Disorder (PTSD)
Brief Title: Randomized, Double-blind, Placebo-Controlled Pilot Study of MDMA-assisted Therapy for PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-9
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: MDMA; Posttraumatic stress disorder; PTSD; Israel; psychotherapy; midomafetamine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Lead in: 125 mg MDMA-assisted therapy (Open-Label) (Experimental): Participants receive open-label MDMA with an initial dose of 125 mg midomafetamine HCl, possibly followed by a supplemental dose of 62.5 mg, during two psychotherapy sessions scheduled 3-5 weeks apart.
  Interventions: Drug: Open-Label Full Dose MDMA-assisted therapy (125 mg); Behavioral: Psychotherapy
- Active placebo dose MDMA-assisted therapy (25 mg) (Placebo Comparator): Participants receive initial dose of 25 mg midomafetamine HCl, possibly followed by a supplemental dose of 12.5 mg, during two psychotherapy sessions scheduled 3-5 weeks apart.
  Interventions: Drug: Active Placebo Dose MDMA-assisted therapy (25 mg); Behavioral: Psychotherapy
- Full dose MDMA-assisted therapy (125 mg) (Experimental): Participants receive initial dose of 125 mg midomafetamine HCl, possibly followed by a supplemental dose of 62.5 mg, during two psychotherapy sessions scheduled 3-5 weeks apart.
  Interventions: Drug: Full Dose MDMA-assisted therapy (125 mg); Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Active Placebo Dose MDMA-assisted therapy (25 mg) — Initial dose of 25 mg midomafetamine HCl administered orally at the start of each of two psychotherapy sessions, possibly followed by a supplemental dose of 12.5 mg 1.5 to 2.5 hours later.
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine; MDMA; midomafetamine HCl
  Arms: Active placebo dose MDMA-assisted therapy (25 mg)
Drug: Full Dose MDMA-assisted therapy (125 mg) — Initial dose of 125 mg midomafetamine HCl administered orally at the start of each of two psychotherapy sessions, possibly followed by a supplemental dose of 62.5 mg 1.5 to 2.5 hours later.
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine; MDMA; midomafetamine HCl
  Arms: Full dose MDMA-assisted therapy (125 mg)
Drug: Open-Label Full Dose MDMA-assisted therapy (125 mg) — Initial dose of 125 mg midomafetamine HCl administered orally at the start of each of two psychotherapy sessions, possibly followed by a supplemental dose of 62.5 mg 1.5 to 2.5 hours later.
  Other Names: 3,4-methylenedioxymethamphetamine; midomafetamine; MDMA; midomafetamine HCl
  Arms: Lead in: 125 mg MDMA-assisted therapy (Open-Label)
Behavioral: Psychotherapy — Non-directive psychotherapy will be conducted throughout the study.
  Other Names: Manualized MDMA-assisted psychotherapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people with chronic, treatment-resistant PTSD.

The main question it aims to answer is: Is there a reduction in PTSD symptoms in people given a low dose of MDMA with therapy versus a high dose of MDMA with therapy?

Researchers will compare two sessions of MDMA-assisted therapy with either 25 mg of MDMA HCl or 125 mg of MDMA HCl in Stage 1.

Participants will undergo preparatory therapy sessions without any study drug, followed by two sessions of MDMA-assisted therapy, each followed by integrative therapy sessions without study drug. Participants who received 25 mg during Stage 1 will be given the option to enroll in Stage 2 and complete two additional open-label MDMA-assisted therapy sessions with the full dose of 125 mg MDMA.

DETAILED DESCRIPTION:
This randomized, double-blind, active placebo-controlled Phase 2 pilot study investigated the safety and efficacy of MDMA-assisted psychotherapy in 10 people with chronic, treatment-resistant posttraumatic stress disorder (PTSD), comparing the effects of low and full dose MDMA as an adjunct to psychotherapy. The first two subjects were enrolled in the open label full dose lead-in with 125 mg of midomafetamine HCl, followed by a supplemental half-dose of 62.5 mg after 1.5 to 2.5 hours. The remaining eight subjects enrolled in Stage 1 of the study and received either an active placebo dose (low dose of 25 mg midomafetamine HCl with a supplemental half-dose of 12.5 mg) or a fully active dose (125 mg midomafetamine HCl with a supplemental half-dose of 62.5 mg) during two experimental psychotherapy session, each lasting six to eight hours and scheduled three to five weeks apart.

Upon enrollment, subjects met with their therapist team for three preparatory sessions. After each MDMA-assisted psychotherapy session, subjects met with their therapist team for integrative psychotherapy sessions.

The extent of PTSD symptoms was assessed at baseline and two months after the second experimental session using the Clinician Administered PTSD Scale (CAPS) (Blake et al., 1995). Safety measures, vital signs, and a measurement of psychological distress was assessed during all experimental sessions. Blood pressure and heart rate were assessed periodically during each experimental session.

Subjects who enrolled in Stage 1 and received the active placebo had the opportunity to enroll in Stage 2 of the study and complete open-label experimental sessions with the fully active dose of midomafetamine HCl (125 mg and 62.5 mg supplemental) on the same schedule as Stage 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic PTSD with a duration of 6 months or longer.
* Have a CAPS score showing moderate to severe symptoms.
* Had at least one unsuccessful attempt at treatment for PTSD, either with talk therapy or with drugs, or stopped treatment because of inability to tolerate psychotherapy or drug therapy.
* Are at least 18 years old.
* Generally healthy.
* Must sign a medical release for the investigators to communicate directly with their therapist and doctors.
* Are willing to refrain from taking any psychiatric medications during the study period.
* Agree that, one week before the MDMA session, will refrain from taking all below unless with prior approval of research team: herbal supplements, nonprescription medications (with the exception of nonsteroidal anti-inflammatory drugs or acetaminophen, any prescription medications, with the exception of birth control pills, thyroid hormone, or other medications;
* Are willing to follow restrictions and guidelines concerning consumption of food, beverages. and nicotine the night before and just prior to each experimental session.
* Are willing to remain overnight at the study site.
* Are willing to be contacted via telephone for all necessary telephone contacts.
* Must have a negative pregnancy test if able to bear children, and agree to use an effective form of birth control.
* Agree not to participate in any other clinical trial for the duration of this clinical trial, including the follow-up period.
* Are proficient in speaking and reading Hebrew.
* Agree to have all psychotherapy sessions recorded to audio/video.

Exclusion Criteria:

* Are pregnant or nursing, or if they can have children and are not practicing an effective means of birth control.
* Weigh less than 48 kg.
* Are abusing illegal drugs.
* Have used "Ecstasy" (material represented as containing MDMA) more than five times or at least once within 6 months of the MDMA session.
* Are unable to give adequate informed consent.
* Upon review of past and current drugs/medication must not be on or have taken a medication that is exclusionary.
* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2017-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Kotler, Principal Investigator — Beer Yaakov Hospital
Locations (1):
- Beer Yaakov Hospital, Be’er Ya‘aqov, Israel

REFERENCES:
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Derived] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Derived] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Derived] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through printed ads, internet ads, referrals from other psychiatrists, psychotherapists or physicians, through the Israeli Defense Forces (IDF) and through word of mouth.
Groups:
- Open-Label: 125 mg MDMA-assisted Therapy: Open label: Participants receive initial dose of 125 mg midomafetamine HCl possibly followed by a supplemental dose of 62.5 mg during two psychotherapy sessions.
- Blinded: Full Dose MDMA-assisted Therapy: Participants receive initial dose of 125 mg midomafetamine HCl possibly followed by a supplemental dose of 62.5 mg during two psychotherapy sessions scheduled 3-5 weeks apart.
- Blinded: Active Placebo Dose MDMA-assisted Therapy: Participants receive initial doses of 25 mg midomafetamine HCl possibly followed by a supplemental dose of 12.5 mg during two psychotherapy sessions scheduled 3-5 weeks apart.
Period: Stage 1
Arm/Group | Open-Label: 125 mg MDMA-assisted Therapy | Blinded: Full Dose MDMA-assisted Therapy | Blinded: Active Placebo Dose MDMA-assisted Therapy
Started | 2 | 5 | 3
Completed (Stage 1 Completion) | 2 | 5 | 3
Not Completed | 0 | 0 | 0
Period: Stage 2
Arm/Group | Open-Label: 125 mg MDMA-assisted Therapy | Blinded: Full Dose MDMA-assisted Therapy | Blinded: Active Placebo Dose MDMA-assisted Therapy
Started | 0 | 0 | 2
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 0
Period: 12 Month Follow-Up
Arm/Group | Open-Label: 125 mg MDMA-assisted Therapy | Blinded: Full Dose MDMA-assisted Therapy | Blinded: Active Placebo Dose MDMA-assisted Therapy
Started | 2 | 5 | 3
Completed | 2 | 5 | 2
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lead in: 125 mg MDMA (Open Label) and Psychotherapy: Participants receive open MDMA with an initial dose of 125 mg MDMA possibly followed by a supplemental dose of 62.5 mg during two psychotherapy sessions.
- Full Dose MDMA (125 mg) and Psychotherapy: Participants receive initial dose of 125 mg MDMA possibly followed by a supplemental dose of 62.5 mg during two psychotherapy sessions scheduled 3-5 weeks apart.
- Active Placebo Dose MDMA (25 mg) and Psychotherapy: Participants receive initial doses of 25 mg MDMA possibly followed by a supplemental dose of 12.5 mg during two psychotherapy sessions scheduled 3-5 weeks apart.
- Total: Total of all reporting groups
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Total
Number analyzed (Participants) | 2 | 5 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (19.72) | 35.1 (10.21) | 38.5 (8.68) | 37.2 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 4
  Male | 1 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White/Caucasian | 2 | 5 | 2 | 9
  Ethnicity: Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Administered PTSD Scale (CAPS-IV) Total Score From Baseline to End of Stage 1
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-IV. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline to 1-Month Post Experimental Session 2 (End of Stage 1)
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lead in: 125 mg MDMA (Open Label) and Psychotherapy: Open label: Participants receive open-label MDMA with initial dose of 125 mg MDMA possibly followed by a supplemental dose of 62.5 mg during two psychotherapy sessions.
- Active Placebo Dose MDMA (25 mg) and Psychotherapy: Participants receive initial dose of 25 mg MDMA possibly followed by a supplemental dose of 12.5 mg during two psychotherapy sessions scheduled 3-5 weeks apart.
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 3 | 5
score on a scale | -42.0 (9.90) | -9.0 (15.62) | -34.6 (16.29)

2. Secondary Outcome: Change in Clinical Administered PTSD Scale (CAPS-IV) Total Score From Baseline to End of Stage 2
Description: as for outcome 1
Time Frame: Baseline to End of Stage 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stage 2 Open-Label Crossover 125 mg MDMA-assisted Therapy: Stage 1: Participants receive initial dose of 25 mg midomafetamine HCl possibly followed by a supplemental dose of 12.5 mg during two psychotherapy sessions scheduled 3-5 weeks apart.
  Stage 2: Participants crossover to receive two open-label sessions of MDMA-assisted therapy with 125 mg midomafetamine HCl followed by a supplemental dose of 62.5 mg.
Arm/Group | Stage 2 Open-Label Crossover 125 mg MDMA-assisted Therapy
Number analyzed (Participants) | 2
score on a scale | -23.0 (15.56)

3. Secondary Outcome: Change in Clinical Administered PTSD Scale (CAPS-IV) Total Score From Baseline to Long-Term Follow-Up
Description: as for outcome 1
Time Frame: Baseline to 12 months post-final experimental session
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 2 | 5
score on a scale | -39.0 (14.14) | -34.5 (20.51) | -48.8 (20.39)

4. Secondary Outcome: Change in Beck Depression Inventory (BDI-II) Total Scores From Baseline to End of Stage 1
Description: Validated self-report measure of symptoms of depression. The BDI-II total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depressive symptoms. The BDI-II is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63.
Time Frame: Baseline to 1-Month Post Experimental Session 2 (End of Stage 1)
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 3 | 5
score on a scale | -17.0 (2.83) | 0.3 (4.73) | -17.0 (12.59)

5. Secondary Outcome: Change in Beck Depression Inventory (BDI-II) Total Score From Baseline to End of Stage 2
Description: as for outcome 4
Time Frame: Baseline to End of Stage 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Open-Label Crossover 125 mg MDMA-assisted Therapy
Number analyzed (Participants) | 2
score on a scale | -6.5 (4.95)

6. Secondary Outcome: Change in Beck Depression Inventory (BDI-II) Total Scores From Baseline to Long-Term Follow-Up
Description: as for outcome 4
Time Frame: Baseline to 12 month post-final experimental session
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 2 | 5
score on a scale | -17.0 (5.66) | -3.5 (4.95) | -18.4 (11.10)

7. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Scale From Baseline to End of Stage 1
Description: The Global Assessment of Functioning (GAF) Scale is a numeric scale ranging from 0 through 100 that is used by mental health clinicians and physicians to subjectively rate the social, occupational, and psychological functioning of adults. Higher scores indicate better functioning.
Time Frame: Baseline to 1-Month Post 2nd Experimental Session (End of Stage 1)
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 3 | 5
score on a scale | 15.0 (21.21) | -2.3 (8.74) | 18.2 (11.14)

8. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Scale From Baseline to End of Stage 2
Description: as for outcome 7
Time Frame: Baseline to End of Stage 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Open-Label Crossover 125 mg MDMA-assisted Therapy
Number analyzed (Participants) | 2
score on a scale | 8.0 (9.90)

9. Secondary Outcome: Change in Global Assessment of Functioning (GAF) Scale From Baseline to Long-Term Follow-Up
Description: as for outcome 7
Time Frame: Baseline to 12 months post-final experimental session
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 2 | 5
score on a scale | 5 (7.07) | -1.5 (0.71) | 26.6 (10.33)

10. Secondary Outcome: Change in Posttraumatic Stress Diagnostic Scale (PDS) Symptom Severity Score From Baseline to End of Stage 1
Description: The Posttraumatic Stress Diagnostic Scale (PDS) is a 49-item self-report instrument designed to aid in the diagnosis of PTSD. Responses to 17 symptom items are made on a 4 point scale ranging from 0 (not at all) to 3 (five or more times per week). The symptom items are summed to calculate the symptom severity score which ranges from 0 to 51, with higher scores indicating more severe PTSD symptoms.
Time Frame: Baseline to 1-Month Post 2nd Experimental Session (End of Stage 1)
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 3 | 5
score on a scale | -19.0 (5.66) | 1.3 (13.43) | -17.4 (9.91)

11. Secondary Outcome: Change in Posttraumatic Stress Diagnostic Scale (PDS) Symptom Severity Score From Baseline to End of Stage 2
Description: as for outcome 10
Time Frame: Baseline to End of Stage 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Open-Label Crossover 125 mg MDMA-assisted Therapy
Number analyzed (Participants) | 2
score on a scale | -11.5 (10.61)

12. Secondary Outcome: Change in Posttraumatic Stress Diagnostic Scale (PDS) Symptom Severity Score From Baseline to Long-Term Follow-Up
Description: as for outcome 10
Time Frame: Baseline to 12 months post-final experimental session
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 2 | 5
score on a scale | -23.0 (0) | -10 (9.90) | -20.4 (12.70)

13. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) From Baseline to End of Stage 1
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances. It is comprised of 18 items that yield seven component scores. Component scores are summed to create a total score. Total scores range from 0 (better) to 21 (worse), with higher scores indicating poor sleep quality.
Time Frame: Baseline to 1-Month Post 2nd Experimental Session (End of Stage 1)
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 3 | 5
score on a scale | -7.5 (6.36) | 1.0 (5.29) | -1.8 (4.44)

14. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) From Baseline to End of Stage 2
Description: as for outcome 13
Time Frame: Baseline to End of Stage 2
Population: Crossover set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Open-Label Crossover 125 mg MDMA-assisted Therapy
Number analyzed (Participants) | 2
score on a scale | -3.5 (3.54)

15. Secondary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) From Baseline to Long-Term Follow-Up
Description: as for outcome 13
Time Frame: Baseline to 12 months post-final experimental session
Population: Intent-to-Treat set (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lead in: 125 mg MDMA (Open Label) and Psychotherapy | Active Placebo Dose MDMA (25 mg) and Psychotherapy | Full Dose MDMA (125 mg) and Psychotherapy
Number analyzed (Participants) | 2 | 2 | 5
score on a scale | -3.5 (3.54) | -2.0 (4.24) | -2.2 (5.40)

ADVERSE EVENTS:
Time Frame: From baseline to study completion (approximately 18 months)
Groups:
- Lead In Open-Label: 125 mg MDMA-assisted Therapy: Participants receive initial dose of 125 mg midomafetamine HCl possibly followed by a supplemental dose of 62.5 mg during two therapy sessions.
- Blinded Full Dose MDMA-assisted Therapy (125 mg) (Stage 1): Participants receive initial dose of 125 mg midomafetamine HCl possibly followed by a supplemental dose of 62.5 mg during two therapy sessions scheduled 3-5 weeks apart.
- Blinded Active Placebo MDMA-assisted Therapy (Stage 1): Participants receive initial dose of 25 mg midomafetamine HCl possibly followed by a supplemental dose of 12.5 mg during two therapy sessions scheduled 3-5 weeks apart.
- Open-Label Full Dose MDMA-assisted Therapy (125 mg) (Stage 2): Stage 1 activate placebo dose participants receive initial dose of 125 mg midomafetamine HCl possibly followed by a supplemental dose of 62.5 mg during two therapy sessions scheduled 3-5 weeks apart.
- 12 Month Follow-Up: Open-Label Full Dose Lead-In; 12 Month Follow-Up: Blinded Full Dose; 12 Month Follow-Up: Active Placebo Dose: Includes Adverse Events that start on or after the day after end of Stage 1 for subject who did not cross over to Stage 2 or end of Stage 2 through the end of the study.
- SRRs: Full Dose; SRRs: Active Placebo: Spontaneously reported reactions (SRRs) during blinded experimental sessions and 7 days after.
Arm/Group | Lead In Open-Label: 125 mg MDMA-assisted Therapy | Blinded Full Dose MDMA-assisted Therapy (125 mg) (Stage 1) | Blinded Active Placebo MDMA-assisted Therapy (Stage 1) | Open-Label Full Dose MDMA-assisted Therapy (125 mg) (Stage 2) | 12 Month Follow-Up: Open-Label Full Dose Lead-In | 12 Month Follow-Up: Blinded Full Dose | 12 Month Follow-Up: Active Placebo Dose | SRRs: Full Dose | SRRs: Active Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/3 | 0/2 | 0/2 | 0/5 | 0/2 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/3 | 0/2 | 0/2 | 0/5 | 0/2 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 4/5 | 1/3 | 2/2 | 0/2 | 1/5 | 0/3 | 5/5 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lead In Open-Label: 125 mg MDMA-assisted Therapy (N=2) | Blinded Full Dose MDMA-assisted Therapy (125 mg) (Stage 1) (N=5) | Blinded Active Placebo MDMA-assisted Therapy (Stage 1) (N=3) | Open-Label Full Dose MDMA-assisted Therapy (125 mg) (Stage 2) (N=2) | 12 Month Follow-Up: Open-Label Full Dose Lead-In (N=2) | 12 Month Follow-Up: Blinded Full Dose (N=5) | 12 Month Follow-Up: Active Placebo Dose (N=3) | SRRs: Full Dose (N=5) | SRRs: Active Placebo (N=3)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Posttraumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exposure to violent event (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drowsiness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Heavy legs (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Jaw Clenching, Tight Jaw (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lack of Appetite (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Low mood (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Muscle tension (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Need more sleep (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Perspiration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weakness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT01689740/Prot_004.pdf
  • Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT01689740/SAP_001.pdf
  • Informed Consent Form (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT01689740/ICF_003.pdf